CLINICAL TRIAL: NCT05172466
Title: Sensation, Motion, and Quality of Life on Natalizumab and Off Natalizumab
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack on enrollment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Laura Tabacof, Principal Investigator, Research Instructor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY-20-02068
Record Dates: First submitted 2021-11-22; First posted 2021-12-29 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Relapsing-remitting Multiple Sclerosis (RRMS)
Keywords: Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Mobile Applications; Natalizumab; Smartphone
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BeCare application (Experimental): individuals with relapsing-remitting MS (RRMS) on Natalizumab therapy
  Interventions: Device: BeCare application

INTERVENTIONS:
Device: BeCare application — Participants will complete activities on the application 3 times a week for 2 weeks when they first join the study. They will then attend 4 in-person visits where they complete clinical and application based assessments. Activities are clearly marked in the application and participants are assigned specific assessments by the study team. The application analyzes user input during each evaluation to provide an outcome measure for that assessment.

SUMMARY:
The goal of this proposal is to use the BeCare App to (1) determine changes in "Feel Good Effect", or "Restoring Physiologic Homeostasis(RPH)"for individuals with relapsing-remitting MS (RRMS) before and after starting Natalizumab therapy and (2) Compare BeCare-derived with clinically-derived performance metrics.

DETAILED DESCRIPTION:
Relapsing-remitting Multiple sclerosis (MS) is a chronic and often disabling disease that has been linked to a wide range of symptoms. Traditionally, MS-related symptoms have been evaluated using functional assessments such as the Kurtzke Expanded Disability Status Scale (EDSS) and the Timed Up and Go (TUG) Test. Detecting subtle changes in kinetic function is a key component in the monitoring and measuring of disease progression as well as predicting outcomes in MS. The BeCare Link mobile application provides validated, quantitative measurements of physical and cognitive functioning to give high precision measurement of disease status and treatment outcomes. Natalizumab is an effective drug that modulates immunity and inflammatory burden over time. While clinical outcomes in controlled clinical trials have shown that Natalizumab results in a reduction in disease progression on the EDSS, there is an often-referenced anecdotal effect reported by patients treated with Tysabri that they feel closer to their overall pre-MS sense of well-being, such as improved speed of cognition, reduced fatigue, and swifter motor and sensory function. This was named "Feel Good Effect", or "Restoring Physiologic Homeostasis(RPH)". Quantification of this effect has not been addressed previously.

This is a prospective single-center study. The goal of this proposal is to use the BeCare App to (1) determine changes in RPH for individuals with relapsing-remitting MS (RRMS) before and after starting Natalizumab therapy and (2) Compare BeCare-derived with clinically-derived performance metrics. Changes in RPH will be determined by pre/post differences in EDSS scores and self-reported questions regarding mood, quality of life, function and participation. The hypothesis is that Natalizumab will be associated with a significant improvement in RPH that will be quantifiable through the use of the BeCare App. The aim is to enroll 20 subjects, recruited from Mount Sinai MS clinic or self referred by contacting the study contact information posted on ClinicalTrials.gov. Individuals included will be of ages between 18 and 60 years with diagnosed RRMS (relapsing-remitting MS) who were prescribed Tysabri (Natalizumab) by their physician. Potential participants will contact the coordinator via phone call or e-mail and will be consented. After consent, participants will download the BeCare mobile application and be instructed to perform tasks on the app at their home 3 times per week for 2 weeks. Once they schedule their first Tysabri infusion, participants will come to 4 in-person study visits. At each visit, they will perform multiple application-based and clinically-based assessments. The entire study protocol will last up to 32 weeks, including follow up. All procedures of this trial are non-invasive and imply minimal risk. All study procedures involve clinical assessments performed routinely as part of their clinical care. Risks involve loss of private information and falling during the study tasks. Drug administration is not part of the trial, and it will be given as part of clinical care.

Each assessment is performed by the clinician once and the application once. These assessments include the Expanded Disability Status Scale (EDSS), Timed Up and Go (TUG), Tap Task, Path Test, Transcription Test, Timed 25-foot walk, Coded Message Cognitive Test, Six-minute walk test, Contrast sensitivity test, Arm elevation test, Memory test, Vibration test, and the Stroop color and word test (SCWT), 9 Whole Peg Test, Red Saturation Test and self-reported mood, quality of life, function, and participation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis: RRMS (relapsing-remitting MS) or Multiple Sclerosis (Clinically Isolated Syndrome [CIS], Primary Progressive [PPMS], Secondary Progressive [SPMS)
* Prescribed Tysabri (Natalizumab) or any other MS medication
* Natalizumab/Tysabri-naïve
* Ages 18-60
* Access to a smartphone* *In case a participant is ineligible due to lack of access to the technology, the study team will loan a tablet to participants for the duration of the study, free of charge. Participants will not be responsible for losing or damaging the device.

Exclusion Criteria:

* Inability to perform 5 or more of the BeCare App tasks independently
* EDSS >6.5
* Corrective Visual Acuity lower than 20/200
* Any chronic illness that has not been stable for at least six months (medication changes during the past year for that condition are not exclusionary)
* Malignancy/previous chemotherapy treatment for neoplastic disease
* Untreated or unstable major depression or bipolar disease
* Clinical diagnosis: SPMS (Secondary-progressive multiple sclerosis) or PPMS (primary-progressive MS) 8. Acute COVID-19 infection with persisting symptoms for the last 6 weeks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
The Expanded Disability Status Scale (EDSS) | Week 0 to 4
  The EDSS is a method of quantifying disability in MS and monitoring changes in the level of disability over time. EDSS steps 1.0 to 4.5 refer to people with MS who are able to walk without any aid and is based on measures of impairment in eight functional systems (FS): (1) pyramidal - muscle weakness or difficulty moving limbs;(subscale 0-6); (2) cerebellar - ataxia, loss of balance, coordination or tremor (subscale 0-5); (3) brainstem - problems with speech, swallowing, and nystagmus (subscale 0-5); (4) sensory - numbness or loss of sensations (subscale 0-6); (5) bowel and bladder function subscale (0-5); (6) visual function - problems with sight (subscale 0-6); (7) cerebral functions - problems with thinking and memory (subscale 0-5); (8) other (subscale 0-1). A functional system (FS) represents a network of neurons in the brain with responsibility for particular tasks. The total scale from 1 - 10, with higher score indicting more severe disability.
The Expanded Disability Status Scale (EDSS) | Week 1-6
  The EDSS is a method of quantifying disability in MS and monitoring changes in the level of disability over time. EDSS steps 1.0 to 4.5 refer to people with MS who are able to walk without any aid and is based on measures of impairment in eight functional systems (FS): (1) pyramidal - muscle weakness or difficulty moving limbs;(subscale 0-6); (2) cerebellar - ataxia, loss of balance, coordination or tremor (subscale 0-5); (3) brainstem - problems with speech, swallowing, and nystagmus (subscale 0-5); (4) sensory - numbness or loss of sensations (subscale 0-6); (5) bowel and bladder function subscale (0-5); (6) visual function - problems with sight (subscale 0-6); (7) cerebral functions - problems with thinking and memory (subscale 0-5); (8) other (subscale 0-1). A functional system (FS) represents a network of neurons in the brain with responsibility for particular tasks. The total scale from 1 - 10, with higher score indicting more severe disability.
The Expanded Disability Status Scale (EDSS) | Week 12-18
  The EDSS is a method of quantifying disability in MS and monitoring changes in the level of disability over time. EDSS steps 1.0 to 4.5 refer to people with MS who are able to walk without any aid and is based on measures of impairment in eight functional systems (FS): (1) pyramidal - muscle weakness or difficulty moving limbs;(subscale 0-6); (2) cerebellar - ataxia, loss of balance, coordination or tremor (subscale 0-5); (3) brainstem - problems with speech, swallowing, and nystagmus (subscale 0-5); (4) sensory - numbness or loss of sensations (subscale 0-6); (5) bowel and bladder function subscale (0-5); (6) visual function - problems with sight (subscale 0-6); (7) cerebral functions - problems with thinking and memory (subscale 0-5); (8) other (subscale 0-1). A functional system (FS) represents a network of neurons in the brain with responsibility for particular tasks. The total scale from 1 - 10, with higher score indicting more severe disability.
The Expanded Disability Status Scale (EDSS) | Week 24-32
  The EDSS is a method of quantifying disability in MS and monitoring changes in the level of disability over time. EDSS steps 1.0 to 4.5 refer to people with MS who are able to walk without any aid and is based on measures of impairment in eight functional systems (FS): (1) pyramidal - muscle weakness or difficulty moving limbs;(subscale 0-6); (2) cerebellar - ataxia, loss of balance, coordination or tremor (subscale 0-5); (3) brainstem - problems with speech, swallowing, and nystagmus (subscale 0-5); (4) sensory - numbness or loss of sensations (subscale 0-6); (5) bowel and bladder function subscale (0-5); (6) visual function - problems with sight (subscale 0-6); (7) cerebral functions - problems with thinking and memory (subscale 0-5); (8) other (subscale 0-1). A functional system (FS) represents a network of neurons in the brain with responsibility for particular tasks. The total scale from 1 - 10, with higher score indicting more severe disability.

SECONDARY OUTCOMES:
Application Based - Timed Up and Go (TUG) | Week 0 to 4
  A validated assessment of functional mobility. The participant is seated in a regular chair with no chair arm-rests. The participant will hold their mobile device in their hand, select the task on the application, and will perform the task without external cue. At the start of the test subjects will stand and walk to a mark three meters from where their feet are placed when sitting, turn 180 degrees, walk back to the chair, and sit to finish. The test result is recorded as the time from start to finish, with a shorter time indicating a lower level of impairment.
Application Based - Timed Up and Go (TUG) | Week 1-6
  A validated assessment of functional mobility. The participant is seated in a regular chair with no chair arm-rests. The participant will hold their mobile device in their hand, select the task on the application, and will perform the task without external cue. At the start of the test subjects will stand and walk to a mark three meters from where their feet are placed when sitting, turn 180 degrees, walk back to the chair, and sit to finish. The test result is recorded as the time from start to finish, with a shorter time indicating a lower level of impairment.
Application Based - Timed Up and Go (TUG) | Week 12-18
  A validated assessment of functional mobility. The participant is seated in a regular chair with no chair arm-rests. The participant will hold their mobile device in their hand, select the task on the application, and will perform the task without external cue. At the start of the test subjects will stand and walk to a mark three meters from where their feet are placed when sitting, turn 180 degrees, walk back to the chair, and sit to finish. The test result is recorded as the time from start to finish, with a shorter time indicating a lower level of impairment.
Application Based - Timed Up and Go (TUG) | Week 24-32
  A validated assessment of functional mobility. The participant is seated in a regular chair with no chair arm-rests. The participant will hold their mobile device in their hand, select the task on the application, and will perform the task without external cue. At the start of the test subjects will stand and walk to a mark three meters from where their feet are placed when sitting, turn 180 degrees, walk back to the chair, and sit to finish. The test result is recorded as the time from start to finish, with a shorter time indicating a lower level of impairment.
Application Based - Tap Task | Week 0 to 4
  Participants will be presented with a game on their mobile phone that requires them to tap a designated spot as frequently as possible for 10 seconds. The phone will record the number of taps, the regularity of their spacing, and any consistent change over time (fatigue). The test will be repeated 3 times. These measures will be used to make a determination on level of impairment. Higher quantity of taps, more regular spacing, and limited change over time is indicative of a lower level of impairment.
Application Based - Tap Task | Week 1-6
  Participants will be presented with a game on their mobile phone that requires them to tap a designated spot as frequently as possible for 10 seconds. The phone will record the number of taps, the regularity of their spacing, and any consistent change over time (fatigue). The test will be repeated 3 times. These measures will be used to make a determination on level of impairment. Higher quantity of taps, more regular spacing, and limited change over time is indicative of a lower level of impairment.
Application Based - Tap Task | Week 12-18
  Participants will be presented with a game on their mobile phone that requires them to tap a designated spot as frequently as possible for 10 seconds. The phone will record the number of taps, the regularity of their spacing, and any consistent change over time (fatigue). The test will be repeated 3 times. These measures will be used to make a determination on level of impairment. Higher quantity of taps, more regular spacing, and limited change over time is indicative of a lower level of impairment.
Application Based - Tap Task | Week 24-32
  Participants will be presented with a game on their mobile phone that requires them to tap a designated spot as frequently as possible for 10 seconds. The phone will record the number of taps, the regularity of their spacing, and any consistent change over time (fatigue). The test will be repeated 3 times. These measures will be used to make a determination on level of impairment. Higher quantity of taps, more regular spacing, and limited change over time is indicative of a lower level of impairment.
Application Based - Path Test | Week 0 to 4
  This task asks participants to move an object in the application with their index finger on such that it stays within the boundaries of a moving path. The App will measure deviations outside the path as well as circumstances in which these deviations occur. The test will be repeated 3 times on each side. A lower number of deviations is indicative of a lower level of impairment.
Application Based - Path Test | Week 1-6
  This task asks participants to move an object in the application with their index finger on such that it stays within the boundaries of a moving path. The App will measure deviations outside the path as well as circumstances in which these deviations occur. The test will be repeated 3 times on each side. A lower number of deviations is indicative of a lower level of impairment.
Application Based - Path Test | Week 12-18
  This task asks participants to move an object in the application with their index finger on such that it stays within the boundaries of a moving path. The App will measure deviations outside the path as well as circumstances in which these deviations occur. The test will be repeated 3 times on each side. A lower number of deviations is indicative of a lower level of impairment.
Application Based - Path Test | Week 24-32
  This task asks participants to move an object in the application with their index finger on such that it stays within the boundaries of a moving path. The App will measure deviations outside the path as well as circumstances in which these deviations occur. The test will be repeated 3 times on each side. A lower number of deviations is indicative of a lower level of impairment.
Application Based - Transcription test | Week 0 to 4
  In this test the subject is given a short auditory phrase and then must type that phrase using a virtual keyboard. The time to complete typing the phrase as well as the time-interval and time-variance between keystrokes is compiled. To control for fine motor function, the virtual keyboard records the time and variance for tapping a series of keys that spontaneously change color (white background to green for example), which is termed the maximal keystroke velocity (strokes/second). A higher maximal keystroke velocity, a lower time-interval, and lower time-variance are associated with a lower level of impairment.
Application Based - Transcription test | Week 1-6
  In this test the subject is given a short auditory phrase and then must type that phrase using a virtual keyboard. The time to complete typing the phrase as well as the time-interval and time-variance between keystrokes is compiled. To control for fine motor function, the virtual keyboard records the time and variance for tapping a series of keys that spontaneously change color (white background to green for example), which is termed the maximal keystroke velocity (strokes/second). A higher maximal keystroke velocity, a lower time-interval, and lower time-variance are associated with a lower level of impairment.
Application Based - Transcription test | Week 12-18
  In this test the subject is given a short auditory phrase and then must type that phrase using a virtual keyboard. The time to complete typing the phrase as well as the time-interval and time-variance between keystrokes is compiled. To control for fine motor function, the virtual keyboard records the time and variance for tapping a series of keys that spontaneously change color (white background to green for example), which is termed the maximal keystroke velocity (strokes/second). A higher maximal keystroke velocity, a lower time-interval, and lower time-variance are associated with a lower level of impairment.
Application Based - Transcription test | Week 24-32
  In this test the subject is given a short auditory phrase and then must type that phrase using a virtual keyboard. The time to complete typing the phrase as well as the time-interval and time-variance between keystrokes is compiled. To control for fine motor function, the virtual keyboard records the time and variance for tapping a series of keys that spontaneously change color (white background to green for example), which is termed the maximal keystroke velocity (strokes/second). A higher maximal keystroke velocity, a lower time-interval, and lower time-variance are associated with a lower level of impairment.
Application Based - Timed 25-foot walk | Week 0 to 4
  At the start of the test, the subject is standing at a mark (typically taped on the floor) and is prepared to walk to the destination mark 25 feet away. The participant holds their phone in their hand, selects the test, and then performs the test without a cue. The Subject then walks as quickly as possible while remaining safe, to the 25-foot mark. The test result is recorded as the time from start to finish. A faster time is indicative of a lower level of impairment.
Application Based - Timed 25-foot walk | Week 1-6
  At the start of the test, the subject is standing at a mark (typically taped on the floor) and is prepared to walk to the destination mark 25 feet away. The participant holds their phone in their hand, selects the test, and then performs the test without a cue. The Subject then walks as quickly as possible while remaining safe, to the 25-foot mark. The test result is recorded as the time from start to finish. A faster time is indicative of a lower level of impairment.
Application Based - Timed 25-foot walk | Week 12-18
  At the start of the test, the subject is standing at a mark (typically taped on the floor) and is prepared to walk to the destination mark 25 feet away. The participant holds their phone in their hand, selects the test, and then performs the test without a cue. The Subject then walks as quickly as possible while remaining safe, to the 25-foot mark. The test result is recorded as the time from start to finish. A faster time is indicative of a lower level of impairment.
Application Based - Timed 25-foot walk | Week 24-32
  At the start of the test, the subject is standing at a mark (typically taped on the floor) and is prepared to walk to the destination mark 25 feet away. The participant holds their phone in their hand, selects the test, and then performs the test without a cue. The Subject then walks as quickly as possible while remaining safe, to the 25-foot mark. The test result is recorded as the time from start to finish. A faster time is indicative of a lower level of impairment.
Application Based - Coded Message Cognitive Test | Week 0 to 4
  Participants are presented with a key where symbols are mapped to a letter or word. The participant is then presented with a list of symbols and asked to convert them to the letter or word. This is a timed test. A faster time is indicative of a lower level of impairment.
Application Based - Coded Message Cognitive Test | Week 1-6
  Participants are presented with a key where symbols are mapped to a letter or word. The participant is then presented with a list of symbols and asked to convert them to the letter or word. This is a timed test. A faster time is indicative of a lower level of impairment.
Application Based - Coded Message Cognitive Test | Week 12-18
  Participants are presented with a key where symbols are mapped to a letter or word. The participant is then presented with a list of symbols and asked to convert them to the letter or word. This is a timed test. A faster time is indicative of a lower level of impairment.
Application Based - Coded Message Cognitive Test | Week 24-32
  Participants are presented with a key where symbols are mapped to a letter or word. The participant is then presented with a list of symbols and asked to convert them to the letter or word. This is a timed test. A faster time is indicative of a lower level of impairment.
Application Based - Six-minute walk test | Week 0 to 4
  Participants are asked to walk at a comfortable pace for 6 minutes while the BeCare application records distance using GPS and records the number of steps taken using the mobile devices accelerometer. A higher distance traveled and number of steps taken is indicative of a lower level of impairment.
Application Based - Six-minute walk test | Week 1-6
  Participants are asked to walk at a comfortable pace for 6 minutes while the BeCare application records distance using GPS and records the number of steps taken using the mobile devices accelerometer. A higher distance traveled and number of steps taken is indicative of a lower level of impairment.
Application Based - Six-minute walk test | Week 12-18
  Participants are asked to walk at a comfortable pace for 6 minutes while the BeCare application records distance using GPS and records the number of steps taken using the mobile devices accelerometer. A higher distance traveled and number of steps taken is indicative of a lower level of impairment.
Application Based - Six-minute walk test | Week 24-32
  Participants are askedParticipants are asked to walk at a comfortable pace for 6 minutes while the BeCare application records distance using GPS and records the number of steps taken using the mobile devices accelerometer. A higher distance traveled and number of steps taken is indicative of a lower level of impairment. to walk at a comfortable pace for 6 minutes while the BeCare application records distance using GPS and records the number of steps taken using the mobile devices accelerometer.
Application Based - Contrast sensitivity test | Week 0 to 4
  For this test the subject is asked to discern or read letters/numerals off a screen with varying contrast sensitivity (grey on grey). Next to each letter/number is a box for them to enter the character/numeral using a virtual keyboard. The number of correct assignments is recorded and reported as a fraction of the total number tested. A greater number of correct assignments is indicative of a lower level of impairment.
Application Based - Contrast sensitivity test | Week 1-6
  For this test the subject is asked to discern or read letters/numerals off a screen with varying contrast sensitivity (grey on grey). Next to each letter/number is a box for them to enter the character/numeral using a virtual keyboard. The number of correct assignments is recorded and reported as a fraction of the total number tested. A greater number of correct assignments is indicative of a lower level of impairment.
Application Based - Contrast sensitivity test | Week 12-18
  For this test the subject is asked to discern or read letters/numerals off a screen with varying contrast sensitivity (grey on grey). Next to each letter/number is a box for them to enter the character/numeral using a virtual keyboard. The number of correct assignments is recorded and reported as a fraction of the total number tested. A greater number of correct assignments is indicative of a lower level of impairment.
Application Based - Contrast sensitivity test | Week 24-32
  For this test the subject is asked to discern or read letters/numerals off a screen with varying contrast sensitivity (grey on grey). Next to each letter/number is a box for them to enter the character/numeral using a virtual keyboard. The number of correct assignments is recorded and reported as a fraction of the total number tested. A greater number of correct assignments is indicative of a lower level of impairment.
Application Based - Arm elevation test | Week 0 to 4
  Participants are asked to hold their mobile device in their dominant hand and then raise their arms to pass the devise to their other hand over the top of their head. This is repeated as fast as possible for 30 seconds. Number of successful passes is measured. A higher number of passes is indicative of lower level of impairment.
Application Based - Arm elevation test | Week 1-6
  Participants are asked to hold their mobile device in their dominant hand and then raise their arms to pass the devise to their other hand over the top of their head. This is repeated as fast as possible for 30 seconds. Number of successful passes is measured. A higher number of passes is indicative of lower level of impairment.
Application Based - Arm elevation test | Week 12-18
  Participants are asked to hold their mobile device in their dominant hand and then raise their arms to pass the devise to their other hand over the top of their head. This is repeated as fast as possible for 30 seconds. Number of successful passes is measured. A higher number of passes is indicative of lower level of impairment.
Application Based - Arm elevation test | Week 24-32
  Participants are asked to hold their mobile device in their dominant hand and then raise their arms to pass the devise to their other hand over the top of their head. This is repeated as fast as possible for 30 seconds. Number of successful passes is measured. A higher number of passes is indicative of lower level of impairment.
Application Based - Memory test | Week 0 to 4
  For this test the subject is presented with 5 animals in 5 colors that appear in boxes in 2 rows, 2 of the boxes with animals are randomly selected and, after 8 seconds, one of the 2 choices are closed. The subject must remember first the animal and color in the box that was closed from the choices that appear, and, on the next round, the subject must remember the previous animal and color from the box that was not presented on the previous round. The choice as to the box that is closed will be mathematically determined to pose the same risk/difficulty for each subject. The number of errors is recorded and the number of correct choices is recorded over 90 seconds. A lower number of errors is indicative of a lower level of impairment.
Application Based - Memory test | Week 1-6
  For this test the subject is presented with 5 animals in 5 colors that appear in boxes in 2 rows, 2 of the boxes with animals are randomly selected and, after 8 seconds, one of the 2 choices are closed. The subject must remember first the animal and color in the box that was closed from the choices that appear, and, on the next round, the subject must remember the previous animal and color from the box that was not presented on the previous round. The choice as to the box that is closed will be mathematically determined to pose the same risk/difficulty for each subject. The number of errors is recorded and the number of correct choices is recorded over 90 seconds. A lower number of errors is indicative of a lower level of impairment.
Application Based - Memory test | Week 12-18
  For this test the subject is presented with 5 animals in 5 colors that appear in boxes in 2 rows, 2 of the boxes with animals are randomly selected and, after 8 seconds, one of the 2 choices are closed. The subject must remember first the animal and color in the box that was closed from the choices that appear, and, on the next round, the subject must remember the previous animal and color from the box that was not presented on the previous round. The choice as to the box that is closed will be mathematically determined to pose the same risk/difficulty for each subject. The number of errors is recorded and the number of correct choices is recorded over 90 seconds. A lower number of errors is indicative of a lower level of impairment.
Application Based - Memory test | Week 24-32
  For this test the subject is presented with 5 animals in 5 colors that appear in boxes in 2 rows, 2 of the boxes with animals are randomly selected and, after 8 seconds, one of the 2 choices are closed. The subject must remember first the animal and color in the box that was closed from the choices that appear, and, on the next round, the subject must remember the previous animal and color from the box that was not presented on the previous round. The choice as to the box that is closed will be mathematically determined to pose the same risk/difficulty for each subject. The number of errors is recorded and the number of correct choices is recorded over 90 seconds. A lower number of errors is indicative of a lower level of impairment.
Application Based - Vibration test | Week 0 to 4
  Participants will be asked to first hold the phone in your right hand and then left hand. The phone will vibrate. The vibration frequency will change several times during the test. Participants will be instructed to hit a box every time to sense a vibration change. Response accuracy will be calculated. A higher level of accuracy is indicative of a lower level of impairment.
Application Based - Vibration test | Week 1-6
  Participants will be asked to first hold the phone in your right hand and then left hand. The phone will vibrate. The vibration frequency will change several times during the test. Participants will be instructed to hit a box every time to sense a vibration change. Response accuracy will be calculated. A higher level of accuracy is indicative of a lower level of impairment.
Application Based - Vibration test | Week 12-18
  Participants will be asked to first hold the phone in your right hand and then left hand. The phone will vibrate. The vibration frequency will change several times during the test. Participants will be instructed to hit a box every time to sense a vibration change. Response accuracy will be calculated. A higher level of accuracy is indicative of a lower level of impairment.
Application Based - Vibration test | Week 24-32
  Participants will be asked to first hold the phone in your right hand and then left hand. The phone will vibrate. The vibration frequency will change several times during the test. Participants will be instructed to hit a box every time to sense a vibration change. Response accuracy will be calculated. A higher level of accuracy is indicative of a lower level of impairment.
Application Based - The Stroop Color and Word Test (SCWT) | Week 0 to 4
  This is a neuropsychological test used to assess the ability to inhibit cognitive interference during simultaneous stimulus processing. Participants will see words written in different colors and will be asked to name the text color. Higher accuracy in naming the text color is indicative of a lower level of impairment.
Application Based - The Stroop Color and Word Test (SCWT) | Week 1-6
  This is a neuropsychological test used to assess the ability to inhibit cognitive interference during simultaneous stimulus processing. Participants will see words written in different colors and will be asked to name the text color. Higher accuracy in naming the text color is indicative of a lower level of impairment.
Application Based - The Stroop Color and Word Test (SCWT) | Week 12-18
  This is a neuropsychological test used to assess the ability to inhibit cognitive interference during simultaneous stimulus processing. Participants will see words written in different colors and will be asked to name the text color. Higher accuracy in naming the text color is indicative of a lower level of impairment.
Application Based - The Stroop Color and Word Test (SCWT) | Week 24-32
  This is a neuropsychological test used to assess the ability to inhibit cognitive interference during simultaneous stimulus processing. Participants will see words written in different colors and will be asked to name the text color. Higher accuracy in naming the text color is indicative of a lower level of impairment.
Application Based - Self-reported mood, quality of life, function, and participation. | Week 0-4
  Questions include: Mood assessment (Angry/Happy/Sad/Frustrated/Tired/Scared); dietary restrictions; employment (Working/Unemployed/Disabled/Cared for a home/student/ retired/ other), frequency of physical exercise (hours/week), presence and severity of cognitive symptoms (concentration, memory, executive function); number of missed work or social events because of MS, presence/absence of other symptoms or events (blurred vision, double vision, altered vision, falls, urinary incontinence).
Application Based - Self-reported mood, quality of life, function, and participation. | Week 1-6
  Questions include: Mood assessment (Angry/Happy/Sad/Frustrated/Tired/Scared); dietary restrictions; employment (Working/Unemployed/Disabled/Cared for a home/student/ retired/ other), frequency of physical exercise (hours/week), presence and severity of cognitive symptoms (concentration, memory, executive function); number of missed work or social events because of MS, presence/absence of other symptoms or events (blurred vision, double vision, altered vision, falls, urinary incontinence).
Application Based - Self-reported mood, quality of life, function, and participation. | Week 12-18
  Questions include: Mood assessment (Angry/Happy/Sad/Frustrated/Tired/Scared); dietary restrictions; employment (Working/Unemployed/Disabled/Cared for a home/student/ retired/ other), frequency of physical exercise (hours/week), presence and severity of cognitive symptoms (concentration, memory, executive function); number of missed work or social events because of MS, presence/absence of other symptoms or events (blurred vision, double vision, altered vision, falls, urinary incontinence).
Application Based - Self-reported mood, quality of life, function, and participation. | Week 24-32
  Questions include: Mood assessment (Angry/Happy/Sad/Frustrated/Tired/Scared); dietary restrictions; employment (Working/Unemployed/Disabled/Cared for a home/student/ retired/ other), frequency of physical exercise (hours/week), presence and severity of cognitive symptoms (concentration, memory, executive function); number of missed work or social events because of MS, presence/absence of other symptoms or events (blurred vision, double vision, altered vision, falls, urinary incontinence).
Clinician Based - The Nine-Hole Peg Test (9HPT) | Week 0 to 4
  The 9HPT is used to measure finger dexterity in patients with various neurological diagnoses. Patients are asked to take the pegs from a container, one by one, and place them into the holes on the board, as quickly as possible. They must then remove the pegs from the holes, one by one, and replace them back into the container. Scores are based on the time taken to complete the test activity, recorded in seconds.
Clinician Based - The Nine-Hole Peg Test (9HPT) | Week 1-6
  The 9HPT is used to measure finger dexterity in patients with various neurological diagnoses. Patients are asked to take the pegs from a container, one by one, and place them into the holes on the board, as quickly as possible. They must then remove the pegs from the holes, one by one, and replace them back into the container. Scores are based on the time taken to complete the test activity, recorded in seconds.
Clinician Based - The Nine-Hole Peg Test (9HPT) | Week 12-18
  The 9HPT is used to measure finger dexterity in patients with various neurological diagnoses. Patients are asked to take the pegs from a container, one by one, and place them into the holes on the board, as quickly as possible. They must then remove the pegs from the holes, one by one, and replace them back into the container. Scores are based on the time taken to complete the test activity, recorded in seconds.
Clinician Based - The Nine-Hole Peg Test (9HPT) | Week 24-32
  The 9HPT is used to measure finger dexterity in patients with various neurological diagnoses. Patients are asked to take the pegs from a container, one by one, and place them into the holes on the board, as quickly as possible. They must then remove the pegs from the holes, one by one, and replace them back into the container. Scores are based on the time taken to complete the test activity, recorded in seconds.
Clinician Based - Red Saturation test | Week 0 to 4
  Red saturation test assesses the integrity of the optic nerve by testing the ocular sensitivity to the red colour. The test is used clinically for the detection of asymmetric optic nerve function and detection of neurophthalmological visual field defects such as hemianopias and quadrantopias.
Clinician Based - Red Saturation test | Week 1-6
  Red saturation test assesses the integrity of the optic nerve by testing the ocular sensitivity to the red colour. The test is used clinically for the detection of asymmetric optic nerve function and detection of neurophthalmological visual field defects such as hemianopias and quadrantopias.
Clinician Based - Red Saturation test | Week 12-18
  Red saturation test assesses the integrity of the optic nerve by testing the ocular sensitivity to the red colour. The test is used clinically for the detection of asymmetric optic nerve function and detection of neurophthalmological visual field defects such as hemianopias and quadrantopias.
Clinician Based - Red Saturation test | Week 24-32
  Red saturation test assesses the integrity of the optic nerve by testing the ocular sensitivity to the red colour. The test is used clinically for the detection of asymmetric optic nerve function and detection of neurophthalmological visual field defects such as hemianopias and quadrantopias.
Clinician Global Impression of Change (CGIC) | Week 0 to 4
  CGIC assess clinician's impression of change on a scale ranging from Much better (1) to Much worse (7).
Clinician Global Impression of Change (CGIC) | Week 1-6
  CGIC assess clinician's impression of change on a scale ranging from Much better (1) to Much worse (7).
Clinician Global Impression of Change (CGIC) | Week 12-18
  CGIC assess clinician's impression of change on a scale ranging from Much better (1) to Much worse (7).
Clinician Global Impression of Change (CGIC) | Week 24-32
  CGIC assess clinician's impression of change on a scale ranging from Much better (1) to Much worse (7).
Patient Global Impression of Change (PGIC ) | Week 0 to 4
  PGIC assess participant's impression of change on a scale ranging from Much better (1) to Much worse (7).
Patient Global Impression of Change (PGIC ) | Week 1-6
  PGIC assess participant's impression of change on a scale ranging from Much better (1) to Much worse (7).
Patient Global Impression of Change (PGIC ) | Week 12-18
  PGIC assess participant's impression of change on a scale ranging from Much better (1) to Much worse (7).
Patient Global Impression of Change (PGIC ) | Week 24-32
  PGIC assess participant's impression of change on a scale ranging from Much better (1) to Much worse (7).
Patient-reported - Multiple Sclerosis - Quality of Life (MS-QOL) | Week 0 to 4
  Multidimensional health-related quality of life measure that combines both generic and MS-specific items. It includes 54 questions generating 12 subscales along with two summary scores, and two additional single-item measures. The 4 subscales are: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health, distress, overall quality of life, and sexual function. Each domain score is converted into a 0-100 score based on the individual item responses, with higher scores indicating better health status or functioning.
Patient-reported - Multiple Sclerosis - Quality of Life (MS-QOL) | Week 1-6
  Multidimensional health-related quality of life measure that combines both generic and MS-specific items. It includes 54 questions generating 12 subscales along with two summary scores, and two additional single-item measures. The 4 subscales are: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health, distress, overall quality of life, and sexual function. Each domain score is converted into a 0-100 score based on the individual item responses, with higher scores indicating better health status or functioning.
Patient-reported - Multiple Sclerosis - Quality of Life (MS-QOL) | Week 12-18
  Multidimensional health-related quality of life measure that combines both generic and MS-specific items. It includes 54 questions generating 12 subscales along with two summary scores, and two additional single-item measures. The 4 subscales are: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health, distress, overall quality of life, and sexual function. Each domain score is converted into a 0-100 score based on the individual item responses, with higher scores indicating better health status or functioning.
Patient-reported - Multiple Sclerosis - Quality of Life (MS-QOL) | Week 24-32
  Multidimensional health-related quality of life measure that combines both generic and MS-specific items. It includes 54 questions generating 12 subscales along with two summary scores, and two additional single-item measures. The 4 subscales are: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health, distress, overall quality of life, and sexual function. Each domain score is converted into a 0-100 score based on the individual item responses, with higher scores indicating better health status or functioning.
Patient Health Questionnaire 9-item (PHQ-9) | Week 0 to 4
  Patient reported instrument that includes questions designed to screen for the presence and severity of major depressive disorder. Full scale from 0-27, with higher score indicating more severe symptoms.
Patient Health Questionnaire 9-item (PHQ-9) | Week 1-6
  Patient reported instrument that includes questions designed to screen for the presence and severity of major depressive disorder. Full scale from 0-27, with higher score indicating more severe symptoms.
Patient Health Questionnaire 9-item (PHQ-9) | Week 12-18
  Patient reported instrument that includes questions designed to screen for the presence and severity of major depressive disorder. Full scale from 0-27, with higher score indicating more severe symptoms.
Patient Health Questionnaire 9-item (PHQ-9) | Week 24-32
  Patient reported instrument that includes questions designed to screen for the presence and severity of major depressive disorder. Full scale from 0-27, with higher score indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Tabacof, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will be kept confidential